CLINICAL TRIAL: NCT05793697
Title: Assessment Of Different Scores In Predicting Outcome In Acute Exacerbation Of Chronic Obstructive Pulmonary Disease Patients In Emergency Department
Brief Title: Assessment Of Different Scores In Predicting Outcome In AECOPD Patients In Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Mostafa Saleh Hussein, Principal investigator, Assiut University
Other Study IDs: different scores in AECOPD
Record Dates: First submitted 2022-11-23; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
evaluate the value of different scores in predicting hospital mortality and Need for MV In patients presented to ED with AECOPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is one of the top three causes of death worldwide, and 90% of deaths occur in low- and middle-income countries.

Acute exacerbation of chronic obstructive pulmonary disease(AECOPD) is defined as an acute change in patient's dyspnea, cough, or sputum beyond normal variability that is sufficient to warrant a change in therapy. AECOPD has a negative effect on the quality of life, admission and readmission rates, and disease progression.

For these reasons, appropriate management of acute exacerbations is recommended by national and international organizations.

Identifying high-risk dying patients on hospital admission helps in triaging them to the required level of care.

The use of early warning scores in follow-up is recommended for the early detection of critically ill patients and the prediction of clinical deterioration. CURB65, BAP65, qSOFA , DECAF and NEWS, which mainly involve mental status, respiratory rate, oxygen saturations, pulse, blood pressure, age, BUN level, etc., can be used to predict AECOPD-associated mortality in ED given the simple structure and data availability.

ELIGIBILITY:
Inclusion Criteria:

* All patient presented to ED with acute exacerbation of COPD.

Exclusion Criteria:

* Patient presented with acute insult affecting other system.
* Patient transferred to other centers.
* Inadequate data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient presented to ED with acute exacerbation of COPD no gender discrimination from 18 years to unlimit age
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2023-05-03 (Estimated); Primary Completion 2024-01-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the value of different scores in predicting hospital mortality | one year
  Assessment Of Different Scores In Predicting Outcome In Acute Exacerbation Of Chronic Obstructive Pulmonary Disease Patients In Emergency Department as DECAF(dyspnea grade V according to eMRCD,esinopenia<0.05x10*9/L,consolidation,acidemia<7.30,atrial fibrillation)
  1=mild,2_3=moderate,4_5=severe can be used to predict AECOPD-associated mortality in ED given the simple structure and data availability.

SECONDARY OUTCOMES:
Value of these scores in predicting need for MV. | one year
  Value of these scores in predicting need for MV in AECOPD patient in ER

CONTACTS AND LOCATIONS:
Overall Officials: reham mo abdelmonem, MD, Study Director — Assiut Uneversity

IPD SHARING:
Plan to Share IPD: Undecided
sharing the result of the study after completion

REFERENCES:
- [Background] Redfern OC, Smith GB, Prytherch DR, Meredith P, Inada-Kim M, Schmidt PE. A Comparison of the Quick Sequential (Sepsis-Related) Organ Failure Assessment Score and the National Early Warning Score in Non-ICU Patients With/Without Infection. Crit Care Med. 2018 Dec;46(12):1923-1933. doi: 10.1097/CCM.0000000000003359. PMID 30130262